CLINICAL TRIAL: NCT03313440
Title: Fiber Intake & Fecal Bulk Enhanced Response
Acronym: Fiber
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wageningen University and Research (Other)
Collaborators: J. Rettenmaier & Sohne GmbH & Co. KG (Unknown)
Responsible Party: Principal Investigator, Diederik Esser, Wageningen University and Research Centre, Wageningen University and Research
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: NL62342.081.17
Record Dates: First submitted 2017-10-06; First posted 2017-10-18 (Actual); Last update posted 2018-07-06 (Actual); Status verified 2018-07

CONDITIONS: Fecal Bulk; Intestinal Health
Keywords: Fibre; diet; fecal bulk

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- high fibre (Experimental): A 10 day increase in daily wheat fiber intake by 18-22 grams/day. Products are provided in boxes that must be consumed each day during the intervention.
  Interventions: Other: High wheat fiber
- low fibre (Experimental): A 10 day control intervention with no additional wheat fibre. Products are provided in boxes that must be consumed each day during the intervention.
  Interventions: Other: Low fiber

INTERVENTIONS:
Other: High wheat fiber — Daily increased fiber intake by 18-22 grams/day. Products are provided in boxes that must be consumed each day during the intervention.
  Arms: high fibre
Other: Low fiber — Control low fiber intervention. Products are provided in boxes that must be consumed each day during the intervention.
  Arms: low fibre

SUMMARY:
Some dietary fibres, including wheat fibres, have shown to increase fecal bulk and improve stool. In previous studies, this effect on fecal bulk was especially studied for intact wheat fibers. Moreover, in most studies, the wheat fiber was offered daily as a single dose in cereals. In this study, we investigate whether an increased intake of extracted wheat fiber, implemented at several time points in a normal daily dietary pattern, can also increase fecal bulk and improve stool frequency and consistency. Here we want to demonstrate that an increase in VITACEL Wheat Fiber intake will enhance fecal bulk, both wet and dry weight and that the enhanced wheat fiber intake will also increase stool frequency and consistency. The study is a double-blind crossover design in which the intervention is based on products enriched by VITACEL Wheat Fiber and control products. Both the control and fiber-enriched intervention will last for 10 days with a wash-out period of at least 4 days. The study will be conducted with 25 healthy male human volunteers in the age between 18-70 years old.Persons will be assigned to the intervention groups. In one of the intervention periods participants receive 'control boxes' with products low in wheat fiber and in the other period they will receive boxes with products enriched with VITACEL Wheat Fiber. During an intervention period of 10 days participants will receive 10 boxes, one for each day. In the last 5 days of the intervention + 1 additional day after the intervention (so in total 6 days), participants will collect their fecal samples to analyse fecal bulk. Daily also a diary has to be kept and questionnaires have to be completed to check compliance to the intervention and assess stool consistency, gut-related complaints.

ELIGIBILITY:
Inclusion Criteria:

* Male
* Apparently healthy (no gastrointestinal complaints, no food allergies and no medication that can influence the outcome of this study
* Age range between 18-70 years old
* BMI between 20 and 30 kg/m2
* Average fiber intake of <23grams per day
* Living in the surrounding area of Wageningen (radius ~20 km)

Exclusion Criteria:

* Any digestive tract disorder that is expected to interfere with this study (e.g. (partial) gastric resection, (hemi)colectomy, Crohn's disease, ulcerative colitis, irritable bowel disease, Coeliac disease)
* Known food allergy (e.g. lactose, gluten, nuts, egg, etc)
* Vegetarians
* Use of pro- or prebiotics
* Use of medication that can interfere with study outcomes (including laxatives, diuretics, antidepressants, codeine or antibiotics)
* Alcohol intake ≥ 40g/day (≥ 3 glasses of beer/wine per day)
* Drug abuse
* Current smokers
* Participation in other clinical trials in the past month

Ages: 18 Years to 70 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2017-10-23 (Actual); Primary Completion 2017-12-01 (Actual); Study Completion 2017-12-01 (Actual)

PRIMARY OUTCOMES:
Fecal bulk | last 5 days of each intervention period
  Wet and dry weight of stool samples in grams

SECONDARY OUTCOMES:
stool consistency | last 5 days of each intervention period
  by Bristol stool chart (type 1-7)
gut-related complaints | last 5 days of each intervention period
  by questionnaires and Visual Analogue Scale (VAS) scores (on a 90mm horizontal line; from no complains (minimal) to serious complains (maximum)). Higher values represent a worse outcome

CONTACTS AND LOCATIONS:
Overall Officials: Nicole de Wit, Dr, Principal Investigator — Stichting Wageningen Research
Locations (1):
- Stichting Wageningen Research, Wageningen, Gelderland, Netherlands

IPD SHARING:
Plan to Share IPD: No